CLINICAL TRIAL: NCT02249650
Title: A Phase I Study to Determine the Maximum Tolerated Dose (MTD) and to Evaluate the Safety, Efficacy and Pharmacokinetics Profiles of TSB-9-W1 in Pre-treated Patients With Metastatic Colorectal Cancer (mCRC).
Brief Title: To Determine the MTD and to Evaluate the Safety, Efficacy and PK Profiles of TSB-9-W1 in Pre-treated Patients With mCRC.
Acronym: TSB-9-W1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Sunpan Biotechnology Development Co., Ltd. (Other)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SUNTSBA20110201
Record Dates: First submitted 2014-09-04; First posted 2014-09-25 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; TSB-9-W1
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TSB-9-W1 cohort (Experimental): TSB-9-W1 200 mg/day (Cohort 1) TSB-9-W1 400 mg/day (Cohort 2) TSB-9-W1 600 mg/day (Cohort 3) TSB-9-W1 800 mg/day (Cohort 4) TSB-9-W1 1000 mg/day (Cohort 5)
  Interventions: Drug: TSB-9-W1

INTERVENTIONS:
Drug: TSB-9-W1 — Product name: TSB-9-W1 Unit dose: 100 mg per capsule Dosage form: Capsule Treatment cycle: A treatment cycle consists of 2-day on-dose oral administering and followed by a 3-day off-dose.
  Other Names: TSB-9-W1(IDS)

SUMMARY:
TSB-9-W1, prepared by Taiwan Sunpan Biotechnology Co., Ltd. (TSB) is a botanical drug and applied patent in the United States (US patent No. 7,138,428 B2), Japan (Patent No.

5441947) and Taiwan (Patent No. I432191 and I282280). The R&D laboratory in TSB is ISO/IEC 17025 certified by Taiwan Accreditation Foundation (TAF) and the laboratory number is 2026.The trade name of TSB-9-W1 is "IDS" in English, the registration number is 01472800 at 2011 by Intellectual Property Office (IPO), Taiwan.

A phase I and pk study to determine the Maximum Tolerated Dose (MTD) and to evaluate the safety and efficacy profiles of TSB-9-W1 in pre-treated patients with metastatic colorectal cancer (mCRC).

there are 5 cohorts and a minimal 2 patients and up to 30 patients are required at phase I.

This is a single arm study. All eligible patients with mCRC will receive TSB-9-W1 treatment.

Each treatment cycle is composed by a contiguous 2-day oral administration and a contiguous 3-day rest. Patient should take the study drug once daily before meal with approximately 250 ml or appropriate amount of water.

DETAILED DESCRIPTION:
Study Design

This study is to establish the MTD of TSB-9-W1 for mCRC patients with a traditional 3+3 dose escalation method.

Study Structure

A dose escalation scenario is designed to determine the MTD according to the DLT.

Dose escalation scale:

The dose levels of investigation product are planned to be administered for determining MTD and DLT.

Dose escalation scenario:

Patients will be enrolled in a cohort of 3 patients for each dose level. Dose escalation will proceed sequentially from the lowest dose cohort. No intra-subject dose escalation is allowed. Each patient's first dose will be at least 3-day apart from the very next patient's first dose.

DLT (except diarrhea) is determined by (NCI-CTCAE) version 4.03 (2010/6/14) defined treatment related toxicity ≥ grade 3 and is worsen from the baseline. Any grade ≥ 3 toxicity (except for diarrhea) is considered a DLT unless there is a clear alternative explanation as to the attribution of the adverse event. Diarrhea event is considered as a DLT if the episode is with NCI-CTCAE Grade of 3 and this event lasts > 3 days despite appropriate supportive cares or if it is a Grade 4 event. Diarrhea event reaches Grade 4 will trigger the patient to withdraw from the study. AEs are evaluated according to the NCI-CTCAE version 4.03 as determined by the investigator to be at least possibly related in causality to the IP administration.

DLT is to be observed during the first 6-treatment cycles (1 cycle = 5 days). If none of the first 3 patients experience DLT, then dose escalation will proceed for the next cohort of patients unless the present dose level is level 5 (1000 mg/day). If 1 of 3 patients develops DLT, the cohort will be expanded to 6 patients (another 3 patients to be added subsequently). If no more than 1 of the 6 patients experiences DLT, then escalation to the next dose level will proceed unless the present dose level is level 5. If more than 1 patient develops DLT in any dose cohort, the dose escalation will be withheld and the prior dose level is considered as the MTD unless present dose level is level 1 (200 mg/day).

Data and Safety Monitoring Board (DSMB) meeting will be held to review safety data prior to each dose escalation

Cut-off criteria Enrolled patients will be treated until disease progression. This study will be ended while either condition below is confirmed.

1. All patients are Disease Progression (PD) or death or loss of follow up.
2. Last treated patient receives 9-month treatment.

Duration of Treatment

TSB-9-W1 in a 5-day treatment cycle until disease progression or study cut-off.

Compensation/reward information

There is no Compensation/reward for subject attend the study.

Results

Primary Endpoint:

MTD and DLTs DCR assessed by RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, age ≥ 20 years old
2. Patient who is eligible and able to participate in the study and accepts to enter the study by signing written informed consent
3. Patient has histologically or cytologically confirmed colorectal adenocarcinoma in stage IV under the Tumor-Node-Metastasis (TNM) staging system
4. Patient must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
5. Patient should have received at least two prior therapies for colorectal cancer (CRC) including oxaliplatin and irinotecan based regimens.
6. Patient should have received at least one of the target therapies for CRC including Cetuximab, Bevacizumab, Panitumumab, Regorafenib, and Ziv-aflibercept.
7. Patient with primary major surgery needs to have elapsed ≥ 2 weeks prior to the planned first study treatment day
8. Patient who has ever received chemotherapy, or immunotherapy, or biologic therapy modalities need to wash-out ≥ 2 weeks prior to the baseline visit
9. Patient who has ever received radiotherapy (including chemoradiation therapy) need to end the course ≥ 2 weeks before baseline visit (palliative radiotherapy can be performed on non-study-related local lesions)
10. Patient's life expectancy ≥ 3 months
11. Within 4 weeks of planned first study treatment day, adequate hematopoietic functions are presented:

    * Total white blood cell (WBC) ≥ 3,000 cells/mm3
    * Absolute neutrophil count (ANC) ≥ 1,500 /mm3
    * Hemoglobin (Hb) ≥ 9.0 g/dL
    * Platelets ≥ 100,000 cells/mm3
12. Within 4 weeks of planned first study treatment day, adequate hepatic and renal functions (AST: aspartate aminotransferase, ALT: alanine aminotransferase, ALP: alkaline phosphatase) are presented:

    * Total bilirubin ≤ 2.0 mg/dL
    * AST ≤ 3 x ULN; liver metastasis patients: AST ≤ 5 x ULN
    * ALT ≤ 3 x ULN; liver metastasis patients: ALT ≤ 5 x ULN
    * ALP ≤ 5 x ULN
    * Creatinine ≤ 1.5 mg/dL
13. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
14. Patient can take food and drug orally
15. Male and female patients should use appropriate contraception method(s) shown below during the study and at least 2 weeks after the end of treatment for female patients.

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

1. Patient who has participated in other investigational studies within 4 weeks prior to the first dose of the study medications
2. Patient has history of another malignancy within 5 years prior to study entry, except curatively treated non-melanoma skin cancer, or cervical cancer in situ
3. Patient with known or suspected hypersensitivity to TSB-9-W1 or its formulation excipients
4. Patient has another severe and/or life-threatening medical disease
5. Patient has immuno-compromised condition, with known autoimmune conditions or human immunodeficiency virus (HIV) seropositivity
6. Patient with active systemic infections, active and clinically significant cardiac diseases, clinically active gastroduodenal ulcers, or medical conditions that may significantly affect adequate absorption of investigational product
7. Patient with known brain metastasis
8. Patient with medical, social or psychological factors interfering with compliance
9. Patient having grade ≥ 3 adverse event (AE) based on National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTCAE) 4.03 except blood total bilirubin, AST, ALT, ALP and creatinine at baseline visit
10. Patient having grade ≥ 1 diarrhea based on NCI-CTCAE 4.03.
11. Patient with a medical history of myocardial infraction in the last 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 3 years
  DLT is to be observed during the first 6-treatment cycles (1 cycle = 5 days). If none of the first 3 patients experience DLT, then dose escalation will proceed for the next cohort of patients unless the present dose level is level 5 (1000 mg/day). If 1 of 3 patients develops DLT, the cohort will be expanded to 6 patients (another 3 patients to be added subsequently). If no more than 1 of the 6 patients experiences DLT, then escalation to the next dose level will proceed unless the present dose level is level 5. If more than 1 patient develops DLT in any dose cohort, the dose escalation will be withheld and the prior dose level is considered as the MTD unless present dose level is level 1 (200 mg/day).
Dose limiting toxicities (DLTs) | 30 days
  DLT (except diarrhea) is determined by (NCI-CTCAE) version 4.03 (2010/6/14) defined treatment related toxicity ≥ grade 3 and is worsen from the baseline. Any grade ≥ 3 toxicity (except for diarrhea) is considered a DLT unless there is a clear alternative explanation as to the attribution of the adverse event. Diarrhea event is considered as a DLT if the episode is with NCI-CTCAE Grade of 3 and this event lasts > 3 days despite appropriate supportive cares or if it is a Grade 4 event. Diarrhea event reaches Grade 4 will trigger the patient to withdraw from the study. AEs are evaluated according to the NCI-CTCAE version 4.03 as determined by the investigator to be at least possibly related in causality to the IP administration.

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Sheng Yang, Bachelor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. J Natl Cancer Inst. 2009 May 20;101(10):708-20. doi: 10.1093/jnci/djp079. Epub 2009 May 12. PMID 19436029
- [Background] Sanoff HK, Sargent DJ, Campbell ME, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Goldberg RM. Five-year data and prognostic factor analysis of oxaliplatin and irinotecan combinations for advanced colorectal cancer: N9741. J Clin Oncol. 2008 Dec 10;26(35):5721-7. doi: 10.1200/JCO.2008.17.7147. Epub 2008 Nov 10. PMID 19001325